CLINICAL TRIAL: NCT03341429
Title: BARI-OPTIMISE: a Double-blinded, Randomised, Placebo-controlled Trial of Liraglutide 3.0 mg in Patients With Poor Weight-loss and a Suboptimal Glucagon-like Peptide-1 Response Following Bariatric Surgery
Brief Title: Evaluation of Liraglutide 3.0mg in Patients With Poor Weight-loss and a Suboptimal Glucagon-like Peptide-1 Response
Acronym: BARIOPTIMISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17/0238
Record Dates: First submitted 2017-10-20; First posted 2017-11-14 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Obesity
Keywords: obesity; GLP-1; liraglutide; diabetes; bariatric surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: This study is a double-blind, randomised, placebo-controlled, two-arm, parallel group, single-site trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator who will conduct the follow-up assessments and the trial subjects will be blinded to participants' allocation and will not be involved in delivering any of the intervention. The statistician conducting the data analysis will be blind to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Daily subcutaneous injection of liraglutide 3.0 mg
  Study dosing of liraglutide:
  Week 1: 0.6 mg once daily Week 2: 1.2 mg once daily Week 3: 1.8 mg once daily Week 4: 2.4 mg once daily Week 5-24: 3.0 mg once daily
  In addition to the daily injection of liraglutide/placebo, participants in both groups will be advised to cut down approximately 500 calories from their usual food intake and to achieve a minimum of 150 minutes per week of physical activity.
  Interventions: Drug: Liraglutide Pen Injector [Saxenda]
- Control (Placebo Comparator): Daily subcutaneous injection of placebo; the same dosage regimen as treatment to be followed.
  In addition to the daily injection of liraglutide/placebo, participants in both groups will be advised to cut down approximately 500 calories from their usual food intake and to achieve a minimum of 150 minutes per week of physical activity.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide Pen Injector [Saxenda] — Daily injection of GLP-1 agonist (liraglutide 3.0 mg) for obese patients presenting poor weight loss (<20%) after bariatric surgery and suboptimal GLP-1 levels.
  Other Names: Saxenda
  Arms: Treatment
Drug: Placebo — Daily subcutaneous injection
  Arms: Control

SUMMARY:
A double-blinded, randomised, placebo-controlled trial of liraglutide 3.0 mg in patients with poor weight-loss and a suboptimal glucagon-like peptide-1 response following bariatric surgery

DETAILED DESCRIPTION:
Subjects with poor weight loss response (<20% of their total weight) following 1 year or more primary gastric bypass or primary sleeve gastrectomy, will be identified from the trial site (University College London Hospital) and participant identification centre (Whittington Hospital) and invited to attend a screening visit. The screening assessment will be undertaken only upon patients providing informed consent to undergo such procedure. Information regarding medical history and concomitant medications will be gathered. In addition, full physical examination, blood test and a meal test will be performed. All female participants of childbearing potential will be tested for pregnancy. Once all data related to the screening visit has been acquired, the investigator will review the participants' eligibility for BARI-OPTIMISE trial. Patients with suboptimal GLP-1 response and fulfilling the inclusion and exclusion criteria will be invited to take part in the trial and asked to sign a second consent form. Assurance of adequate use of contraceptive throughout the trial period will be obtained before a written informed consent is sought. Consented participants will then be asked to attend a baseline visit.

During the baseline visit, data such as body weight, body composition, physical function, physical activity level and health-related quality of life will be collected. Adverse events will be reviewed and a meal test will be repeated. Upon completion of all the baseline procedures, participants will be randomised to receive either subcutaneous injection of liraglutide 3.0 mg or identical placebo for 24 weeks. Participants will be counselled for a calorie-reduced diet and to increase their level of physical activity. Participants will also be taught how to self-administer the treatment (by subcutaneous injection). For safety purpose, subject visits will be carried out at weeks 2, 4, 8, 17 and 24 of the treatment initiation. At all these visits, targeted physical examination will be performed and adverse events will be assessed. End-of-study visit will be over the phone 4 weeks after the end of treatment (i.e. week 28).

ELIGIBILITY:
Inclusion Criteria:

1. Patients, 1 year or more after primary RYGB or primary SG, with poor weight-loss (<20% WL) that is not caused by either a surgical or psychological problem.
2. Adults, 18-64 years inclusive.
3. Suboptimal nutrient-stimulated GLP-1 response assessed by a meal test. Suboptimal active GLP-1 response is defined as a ≤2-fold increase in active GLP-1 circulating levels between time 0 and time 30 minutes.
4. Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control, abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
5. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for trial treatment. NOTE: Subjects are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
6. ≤5 % variation in body weight over preceding 3 months.
7. Fluent in English and able to understand and complete questionnaires.
8. Willing and able to provide written informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Had a surgical procedure other than gastric bypass and sleeve gastrectomy.
2. Pregnant or lactating mothers.
3. Participation in other clinical intervention trial.
4. Lifetime history of suicidal behaviour or severe depression assessed by direct questioning.
5. Clinically significant medical abnormalities (e.g., unstable hypertension, clinically significant ECG abnormalities, liver cirrhosis, AST or ALT > 3x the upper normal limit).
6. Heart rate ≥ 100 beats/minute at screening on two separate measurements.
7. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
8. Renal impairment (estimated glomerular infiltration rate (eGFR <30 ml/min 1.73 m2)
9. Known or suspected hypersensitivity to liraglutide 3.0 mg and placebo or any of the excipients involved in their formulation.
10. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
11. Personal history of pancreatitis.
12. Uncontrolled hypothyroidism or hyperthyroidism.
13. History of stroke, unstable angina, acute coronary syndrome, congestive heart failure New York Heart Association class III-IV within the preceding 12 months.
14. History of arrhythmias.
15. Inflammatory bowel disease.
16. Diabetic gastroparesis.
17. Concomitant GLP-1 receptor agonist usage.
18. Concomitant usage of medications that cause weight gain or weight loss.
19. Concomitant usage of DPPIV-inhibitors.
20. Insulin usage.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
%WL | 24 weeks
  The primary objective of this trial is to compare the efficacy of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration, as an adjunct to diet and exercise, on %WL in participants with poor weight-loss and a sub-optimal active GLP-1 response following primary RYGB or SG at the end of the 24-week treatment period.

SECONDARY OUTCOMES:
%fat | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on % body fat assessed using DXA scanning
Skeletal muscle mass | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on skeletal muscle mass assessed using DXA scanning
Bone mineral density | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on bone mineral density assessed using DXA scanning
Glucose level | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on fasted and meal-stimulated levels of glucose assessed using blood test
Insulin | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on fasted and meal-stimulated levels of insulin assessed using blood test
HbA1c | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on fasted and meal-stimulated levels of HbA1c assessed using blood test
Leptin | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on fasted and meal-stimulated levels of leptin assessed using blood test
Gut Hormones | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on fasted and meal-stimulated levels of gut hormones assessed using blood test
Adipokines | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on fasted and meal-stimulated levels of adipokines assessed using blood test
physical functional assessment | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on physical functioning assessed using the 6-minute walk test (6-MWT)
physical function assessment | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on physical functioning assessed using the sit-to-stand test (STS Test)
physical function assessment | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on physical functioning assessed using hand-grip strength
physical function assessment | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on physical functioning assessed using the Paffenbarger Physical Activity Questionnaire (PPAQ)
HRQoL | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on health related quality of life assessed using an adapted Client Service Receipt Inventory (CSRI)
HRQoL | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on health related quality of life assessed using EuroQol-5D (ED5DEQ-5D)
HRQoL | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on health related quality of life assessed using Impact of weight on quality of life-lite (IWQOL-Lite)
HRQoL | 24 weeks
  To compare the effect of 24-weeks of subcutaneous liraglutide 3.0 mg versus placebo administration as an adjunct to diet and exercise at the end of the 24-week treatment period on health related quality of life assessed using Beck depression inventory (BDI)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Batterham, PhD FRCP, Principal Investigator — UCL
Locations (1):
- UCLH, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participants who agree to, through the consent form, will have some of the study data, any remaining study samples and contact details shared with the ORBiS biobank run by the same Centre for Obesity Research and under the oversight of the same Chief Investigator.
Supporting Information: Study Protocol, ICF
Time Frame: If participants agree by signing the option on the consent form, all of the listed above will be transferred to the ORBiS biobank at the end of the study and will be store there indefinitely, or till further use.

REFERENCES:
- [Background] Lenz M, Richter T, Muhlhauser I. The morbidity and mortality associated with overweight and obesity in adulthood: a systematic review. Dtsch Arztebl Int. 2009 Oct;106(40):641-8. doi: 10.3238/arztebl.2009.0641. Epub 2009 Oct 2. PMID 19890430
- [Background] Fruhbeck G, Toplak H, Woodward E, Yumuk V, Maislos M, Oppert JM; Executive Committee of the European Association for the Study of Obesity. Obesity: the gateway to ill health - an EASO position statement on a rising public health, clinical and scientific challenge in Europe. Obes Facts. 2013;6(2):117-20. doi: 10.1159/000350627. Epub 2013 Apr 3. No abstract available. PMID 23548858
- [Background] Gloy VL, Briel M, Bhatt DL, Kashyap SR, Schauer PR, Mingrone G, Bucher HC, Nordmann AJ. Bariatric surgery versus non-surgical treatment for obesity: a systematic review and meta-analysis of randomised controlled trials. BMJ. 2013 Oct 22;347:f5934. doi: 10.1136/bmj.f5934. PMID 24149519
- [Background] Manning S, Pucci A, Carter NC, Elkalaawy M, Querci G, Magno S, Tamberi A, Finer N, Fiennes AG, Hashemi M, Jenkinson AD, Anselmino M, Santini F, Adamo M, Batterham RL. Early postoperative weight loss predicts maximal weight loss after sleeve gastrectomy and Roux-en-Y gastric bypass. Surg Endosc. 2015 Jun;29(6):1484-91. doi: 10.1007/s00464-014-3829-7. Epub 2014 Sep 20. PMID 25239175
- [Background] Batterham RL, Cummings DE. Mechanisms of Diabetes Improvement Following Bariatric/Metabolic Surgery. Diabetes Care. 2016 Jun;39(6):893-901. doi: 10.2337/dc16-0145. PMID 27222547
- [Background] Jimenez A, Casamitjana R, Flores L, Viaplana J, Corcelles R, Lacy A, Vidal J. Long-term effects of sleeve gastrectomy and Roux-en-Y gastric bypass surgery on type 2 diabetes mellitus in morbidly obese subjects. Ann Surg. 2012 Dec;256(6):1023-9. doi: 10.1097/SLA.0b013e318262ee6b. PMID 22968072
- [Background] Arterburn DE, Bogart A, Sherwood NE, Sidney S, Coleman KJ, Haneuse S, O'Connor PJ, Theis MK, Campos GM, McCulloch D, Selby J. A multisite study of long-term remission and relapse of type 2 diabetes mellitus following gastric bypass. Obes Surg. 2013 Jan;23(1):93-102. doi: 10.1007/s11695-012-0802-1. PMID 23161525
- [Background] Lee MH, Lee WJ, Chong K, Chen JC, Ser KH, Lee YC, Chen SC. Predictors of long-term diabetes remission after metabolic surgery. J Gastrointest Surg. 2015 Jun;19(6):1015-21. doi: 10.1007/s11605-015-2808-1. Epub 2015 Apr 4. PMID 25840670
- [Background] Laurino Neto RM, Herbella FA, Tauil RM, Silva FS, de Lima SE Jr. Comorbidities remission after Roux-en-Y Gastric Bypass for morbid obesity is sustained in a long-term follow-up and correlates with weight regain. Obes Surg. 2012 Oct;22(10):1580-5. doi: 10.1007/s11695-012-0731-z. PMID 22907795
- [Background] Sundbom M, Hedberg J, Marsk R, Boman L, Bylund A, Hedenbro J, Laurenius A, Lundegardh G, Moller P, Olbers T, Ottosson J, Naslund I, Naslund E; Scandinavian Obesity Surgery Registry Study Group. Substantial Decrease in Comorbidity 5 Years After Gastric Bypass: A Population-based Study From the Scandinavian Obesity Surgery Registry. Ann Surg. 2017 Jun;265(6):1166-1171. doi: 10.1097/SLA.0000000000001920. PMID 27429019
- [Background] Lassailly G, Caiazzo R, Buob D, Pigeyre M, Verkindt H, Labreuche J, Raverdy V, Leteurtre E, Dharancy S, Louvet A, Romon M, Duhamel A, Pattou F, Mathurin P. Bariatric Surgery Reduces Features of Nonalcoholic Steatohepatitis in Morbidly Obese Patients. Gastroenterology. 2015 Aug;149(2):379-88; quiz e15-6. doi: 10.1053/j.gastro.2015.04.014. Epub 2015 Apr 25. PMID 25917783
- [Background] Caiazzo R, Lassailly G, Leteurtre E, Baud G, Verkindt H, Raverdy V, Buob D, Pigeyre M, Mathurin P, Pattou F. Roux-en-Y gastric bypass versus adjustable gastric banding to reduce nonalcoholic fatty liver disease: a 5-year controlled longitudinal study. Ann Surg. 2014 Nov;260(5):893-8; discussion 898-9. doi: 10.1097/SLA.0000000000000945. PMID 25379859
- [Background] Mohos E, Jano Z, Richter D, Schmaldienst E, Sandor G, Mohos P, Horzov M, Tornai G, Prager M. Quality of life, weight loss and improvement of co-morbidities after primary and revisional laparoscopic roux Y gastric bypass procedure-comparative match pair study. Obes Surg. 2014 Dec;24(12):2048-54. doi: 10.1007/s11695-014-1314-y. PMID 24913243
- [Background] Raoof M, Naslund I, Rask E, Karlsson J, Sundbom M, Edholm D, Karlsson FA, Svensson F, Szabo E. Health-Related Quality-of-Life (HRQoL) on an Average of 12 Years After Gastric Bypass Surgery. Obes Surg. 2015 Jul;25(7):1119-27. doi: 10.1007/s11695-014-1513-6. PMID 25566743
- [Background] Dirksen C, Jorgensen NB, Bojsen-Moller KN, Kielgast U, Jacobsen SH, Clausen TR, Worm D, Hartmann B, Rehfeld JF, Damgaard M, Madsen JL, Madsbad S, Holst JJ, Hansen DL. Gut hormones, early dumping and resting energy expenditure in patients with good and poor weight loss response after Roux-en-Y gastric bypass. Int J Obes (Lond). 2013 Nov;37(11):1452-9. doi: 10.1038/ijo.2013.15. Epub 2013 Feb 19. PMID 23419600
- [Background] Gerner T, Johansen OE, Olufsen M, Torjesen PA, Tveit A. The post-prandial pattern of gut hormones is related to magnitude of weight-loss following gastric bypass surgery: a case-control study. Scand J Clin Lab Invest. 2014 Apr;74(3):213-8. doi: 10.3109/00365513.2013.877594. Epub 2014 Jan 28. PMID 24472033
- [Background] Blackman A, Foster GD, Zammit G, Rosenberg R, Aronne L, Wadden T, Claudius B, Jensen CB, Mignot E. Effect of liraglutide 3.0 mg in individuals with obesity and moderate or severe obstructive sleep apnea: the SCALE Sleep Apnea randomized clinical trial. Int J Obes (Lond). 2016 Aug;40(8):1310-9. doi: 10.1038/ijo.2016.52. Epub 2016 Mar 23. PMID 27005405
- [Background] Pajecki D, Halpern A, Cercato C, Mancini M, de Cleva R, Santo MA. Short-term use of liraglutide in the management of patients with weight regain after bariatric surgery. Rev Col Bras Cir. 2013 May-Jun;40(3):191-5. doi: 10.1590/s0100-69912013000300005. English, Portuguese. PMID 23912365
- [Derived] Mok J, Adeleke MO, Brown A, Magee CG, Firman C, Makahamadze C, Jassil FC, Marvasti P, Carnemolla A, Devalia K, Fakih N, Elkalaawy M, Pucci A, Jenkinson A, Adamo M, Omar RZ, Batterham RL, Makaronidis J. Safety and Efficacy of Liraglutide, 3.0 mg, Once Daily vs Placebo in Patients With Poor Weight Loss Following Metabolic Surgery: The BARI-OPTIMISE Randomized Clinical Trial. JAMA Surg. 2023 Oct 1;158(10):1003-1011. doi: 10.1001/jamasurg.2023.2930. PMID 37494014